CLINICAL TRIAL: NCT00339365
Title: Promoting Infant Mental Health in Foster Care
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH077329 (NIH); R01MH077329 (NIH); DSIR 84-CTS
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Child Development; Child Behavior Disorders; Reactive Attachment Disorder
Keywords: Infants; Toddlers; Attachment; Maltreatment; Foster Care
MeSH Terms: conditions — Child Behavior Disorders; Reactive Attachment Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Promoting first relationships group
  Interventions: Behavioral: Promoting First Relationships Program
- 2 (Active Comparator): Early education support group
  Interventions: Behavioral: Early Education Support Program

INTERVENTIONS:
Behavioral: Promoting First Relationships Program — Participants assigned to PFR will receive ten weekly home visits that will focus on promoting the development of a secure attachment between foster parents and infants.
  Other Names: PFR
  Arms: 1
Behavioral: Early Education Support Program — EES will consist of three monthly home visits, during which infants will be assessed and referred for additional care if necessary. EES participants will not receive any training.
  Other Names: EES
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of the Promoting First Relationships (PFR) program versus an Early Education Support (EES) program in promoting infant well-being, preventing emotional and behavioral problems, countering developmental delay, and reducing placement instability in young foster care children.

DETAILED DESCRIPTION:
Infants who enter foster care are at risk for developing multiple social and emotional problems later in life. These behavioral issues often result in foster children being placed with multiple different families during their childhoods. In turn, an unstable family life can lead to serious conduct disorders and mental health problems. The infants' loss of their first attachment relationship heightens the risks for developing these problems, even if the quality of care was poor prior to removal. Infants' reactions to this loss, combined with other vulnerabilities, complicate the development of new secure attachments to their foster care families. Garnering a secure attachment relationship between foster parents and foster infants may reduce the infant's risk for developing problematic mental health and conduct issues. PFR is a family therapy intervention focused on aiding foster care parents to cultivate secure attachments with their foster infants. This study will evaluate the effectiveness of the PFR program versus an EES program in promoting attachment security and infant well-being, preventing emotional and behavioral problems, countering developmental delay, and reducing placement instability in young foster care children.

Participants in this single-blind study will be randomly assigned to receive either PFR or EES. Both interventions will be administered by a trained staff member of a community agency. Participants assigned to PFR will receive ten weekly home visits that will focus on promoting the development of a secure attachment between foster parents and infants. EES will consist of three monthly home visits, during which infants will be assessed and referred for additional care if necessary. EES participants will not receive any training. Outcomes will be assessed at 1, 6, and 12 months post-intervention for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Transitioned into foster care, currently within foster care, or from foster care in past three months prior to study entry in Pierce County, WA
* Primary caregiver is foster care provider, kin caregiver, or biological parent

Exclusion Criteria:

* Foster care provider is not English-speaking

Ages: 10 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Toddler Attachment Sort-45 | Measured at Months 1, 6, and 12 post-treatment
Nursing Child Assessment Satellite Training (NCAST) Teaching Scale | Measured at Months 1, 6, and 12 post-treatment
Indicator of Parent-Child Interaction (IPCI) | Measured at Months 1, 6, and 12 post-treatment
Brief Infant-Toddler Social Emotional Assessment | Measured at Months 1, 6, and 12 post-treatment
Bayley Scales of Infant Development, 3rd Edition Screening Test | Measured at baseline and Month 6 post-treatment

SECONDARY OUTCOMES:
Parenting Stress Index/Short Form | Measured at Months 1, 6, and 12 post-treatment
Patient Health Questionnaire (PHQ-9) | Measured at Months 1, 6, and 12 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Susan J. Spieker, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States